CLINICAL TRIAL: NCT01074086
Title: Multicentric Study of GOELAMS Phase I Evaluation of RAD001 in Association With Aracytine and Daunorubicine in AML Treatment in Patients Less Than 65 Years in Relapse More Than One Year After First Complete Remission
Brief Title: Phase I Study in RAD 001 Patients With Relapse AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: RAD 001
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: AML
Keywords: RAD 001 in relapsed AML
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD 001 (Experimental): RAD 001 in day 1 and day 7 from 10 mg to 50 mg
  Interventions: Drug: RAD 001

INTERVENTIONS:
Drug: RAD 001 — RAD 001 in steps of 3 patients from 10mg in day 1 and day 7 to 50 mg
  Other Names: everolimus

SUMMARY:
A phase I clinical study in evaluation of RAD 001 with aracytine and daunorubicine in AML treatment of patients older less than 65 years in relapse

DETAILED DESCRIPTION:
The primary objective of the study is to determinate the maximal tolerate dose and evaluate the toxicity of RAD 001 in patients older less than 65 years in AML relapse in association with a conventional chemotherapy 5Aracytine and Daunorubicine) in an dose escalated phase I study.

ELIGIBILITY:
Inclusion Criteria:

* patients from 18 to 65 years old
* AML in relapse more than 1 year after CR
* inform consent signed

Exclusion Criteria:

* age more than 65
* cardiac insufficiency
* renal insufficiency
* hepatic disease
* other type of AML
* blastic MCL
* HIV positive serology
* other malignancy
* pulmonary infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
maximal dose tolerated | 40 days
  5 steps of RAD 001 doses from 10mg to 50 mg : 3 patienst for each step

SECONDARY OUTCOMES:
Biological study | Day 1 and day 7
  biological study of PI3K/AKT an mTORC1 activation in blast cells
Biological study | Day 1 and Day 7
  concentration mesures of RAD 001 in total blood

CONTACTS AND LOCATIONS:
Overall Officials: Sophie PARK, MD MS, Principal Investigator — French Innovative Leukemia Organisation; Didier BOUSCArY, MD MS, Principal Investigator — French Innovative Leukemia Organisation
Locations (1):
- Sophie Park, Paris, France

REFERENCES:
- [Derived] Park S, Chapuis N, Saint Marcoux F, Recher C, Prebet T, Chevallier P, Cahn JY, Leguay T, Bories P, Witz F, Lamy T, Mayeux P, Lacombe C, Demur C, Tamburini J, Merlat A, Delepine R, Vey N, Dreyfus F, Bene MC, Ifrah N, Bouscary D; GOELAMS (Groupe Ouest Est d'Etude des Leucemies aigues et Autres Maladies du Sang). A phase Ib GOELAMS study of the mTOR inhibitor RAD001 in association with chemotherapy for AML patients in first relapse. Leukemia. 2013 Jul;27(7):1479-86. doi: 10.1038/leu.2013.17. Epub 2013 Jan 16. PMID 23321953